CLINICAL TRIAL: NCT02071498
Title: Effectiveness and Utility of a Virtual Custom Tool to Reduce the Medication Errors of Patients Older Than 65 Years Pluripatologic With Complex Therapeutic Regimens
Brief Title: A Spanish Pillbox App for Elderly Patients Taking Multiple Medications
Acronym: ALICE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Miguel Hernandez de Elche (Other)
Collaborators: Basque Institute for Healthcare Innovation (O+berri), Bilbao, Spain (Unknown); Andalusian Agency for Health Care Quality, Seville, Spain (Unknown); Hospital Universitario Fundación Alcorcón (Other); Castilla-La Mancha Health Service (Other)
Responsible Party: Principal Investigator, José Joaquín Mira, Principal researcher, Universidad Miguel Hernandez de Elche
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: EC11-527; ALICE (Registry Identifier: EC11-527)
Record Dates: First submitted 2014-02-20; First posted 2014-02-26 (Estimated); Last update posted 2014-02-26 (Estimated); Status verified 2014-02

CONDITIONS: Diabetes; Hypertension
Keywords: Pillbox; Non-adherence; Applications; Patient safety; Elderly
MeSH Terms: conditions — Diabetes Mellitus; Hypertension

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pillbox app named ALICE (Experimental): pillbox app for elderly patients taking multiple medications. App was used during three months
  Interventions: Device: Pillbox app named ALICE
- oral and written information (Active Comparator): oral and written information regarding the main risks related to their medications and the most common errors of patients
  Interventions: Other: oral and written information

INTERVENTIONS:
Device: Pillbox app named ALICE — Participants in the experimental group were given a BQ tablet or an iPad with the ALICE app installed and personalised according to the medications they had been prescribed as listed in their medical record
  Arms: Pillbox app named ALICE
Other: oral and written information — oral and written information about the most common errors of patients
  Other Names: information regarding common errors of patients
  Arms: oral and written information

SUMMARY:
Background: Non-adherence and medication errors are common among patients with complex drug regimens. Applications for smartphones and tablets are known to be effective for improving adherence but they have not been tested in elderly patients with such complex chronic conditions, their older age meaning they tend to have less experience with this type of technology.

Objective: to design, implement and evaluate a medication self-management application for elderly patients taking multiple medications called ALICE with the intention of improving adherence and safe medication use.

Methods: A single-blind randomized controlled trial was conducted with a control and an experimental group (N=99) in Spain in 2013. The characteristics of ALICE were specified based on the suggestions of 3 nominal groups with a total of 23 patients and a focus group with 7 professionals. ALICE was designed for Android and iOS and to allow the personalisation of prescriptions and medical advice, showing images of each of the medications (the packaging and the medication itself) together with alerts and multiple reminders for each alert. The randomly subjects in the control group received oral and written information on the safe use of their medications and the experimental group used ALICE for three months. Pre- and post- measures included: rate of missed doses and medication errors reported by patients, Morisky Medication Adherence 4 items Scale scores, level of independence, self-perceived health status and biochemical test results of the patients. In the experimental group, data were also collected on their previous experience with information and communication technologies, their rating of ALICE and their perception of the level of independence they had achieved. The inter-group intervention effects were calculated by univariate linear models and ANOVA, with the pre- to post-intervention differences as the dependent variables.

DETAILED DESCRIPTION:
A tablet-based medication self-management app (called ALICE) was designed to help patients to remember to take all their medications, at the correct doses, distinguish between drugs to avoid confusions, avoid known potential interactions and common errors in use of the medications and know how to properly store the medications. The app design was based on suggestions extracted from 3 nominal groups with a total of 23 patients and a focus group with 7 professionals (3 physicians and 4 pharmacists).

The tablet used was selected on the basis of the need for a device with an at least 7-inch, easy to use touch screen, ensuring that users would only have to follow simple instructions and tap on some icons on the screen. Specifically, the BQ Verne Plus 3G with an LCD Tactile screen was chosen in the case of Android, and an iPad 2 with Wi-Fi + 3G in the case of the iOS.

This study has been approved and financed by the Spanish Ministry of Health, Equality, and Social Policy. The Spanish Research Health Agency (FIS), Independent Clinical Research, project number EC11-527. The Experimental Research Ethics Committee of Miguel Hernández University (DPS-JJM-003-11) approved the trial.

ELIGIBILITY:
Inclusion Criteria:

* Multimorbid patients taking multiple medications
* Over 65 years old, with a Barthel score of more than 60
* Living in their own home
* Able to manage the administration of their medication at home

Exclusion Criteria:

* Refusing to participate in the study
* More than 90 years old

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 99 (Actual)
Dates: Start 2012-06; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
adherence | participants will be followed using ALICE, an expected average of 3 months
  All the participating patients completed a questionnaire (The Morisky Medication Adherence 4 items Scale) to assess the rates of missed doses Number of alerts of the pillbox app that were not dealt

SECONDARY OUTCOMES:
safety medication use | participants will be followed using ALICE, an expected average of 3 months
  avoid most common errors of patients when taking medications (overdoses or confounding pills)

CONTACTS AND LOCATIONS:
Overall Officials: José J Mira, PhD, Principal Investigator — Universidad Miguel Hernández
Locations (1):
- Universidad Miguel Hernández, Elche, Alicante, Spain

REFERENCES:
- [Background] Dayer L, Heldenbrand S, Anderson P, Gubbins PO, Martin BC. Smartphone medication adherence apps: potential benefits to patients and providers. J Am Pharm Assoc (2003). 2013 Mar-Apr;53(2):172-81. doi: 10.1331/JAPhA.2013.12202. PMID 23571625
- [Background] Metlay JP, Cohen A, Polsky D, Kimmel SE, Koppel R, Hennessy S. Medication safety in older adults: home-based practice patterns. J Am Geriatr Soc. 2005 Jun;53(6):976-82. doi: 10.1111/j.1532-5415.2005.53308.x. PMID 15935020
- [Background] Hayakawa M, Uchimura Y, Omae K, Waki K, Fujita H, Ohe K. A smartphone-based medication self-management system with realtime medication monitoring. Appl Clin Inform. 2013 Jan 30;4(1):37-52. doi: 10.4338/ACI-2012-10-RA-0045. Print 2013. PMID 23650486
- [Background] Arsand E, Froisland DH, Skrovseth SO, Chomutare T, Tatara N, Hartvigsen G, Tufano JT. Mobile health applications to assist patients with diabetes: lessons learned and design implications. J Diabetes Sci Technol. 2012 Sep 1;6(5):1197-206. doi: 10.1177/193229681200600525. PMID 23063047
- [Background] Morales Suarez-Varela MT; GEMECOR. [Study on the use of a smart pillbox to improve treatment compliance]. Aten Primaria. 2009 Apr;41(4):185-91. doi: 10.1016/j.aprim.2008.07.003. Epub 2009 Mar 28. Spanish. PMID 19328598
- [Background] Mira JJ, Orozco-Beltran D, Perez-Jover V, Martinez-Jimeno L, Gil-Guillen VF, Carratala-Munuera C, Sanchez-Molla M, Pertusa-Martinez S, Asencio-Aznar A. Physician patient communication failure facilitates medication errors in older polymedicated patients with multiple comorbidities. Fam Pract. 2013 Feb;30(1):56-63. doi: 10.1093/fampra/cms046. Epub 2012 Aug 17. PMID 22904014
- [Derived] Mira JJ, Navarro I, Botella F, Borras F, Nuno-Solinis R, Orozco D, Iglesias-Alonso F, Perez-Perez P, Lorenzo S, Toro N. A Spanish pillbox app for elderly patients taking multiple medications: randomized controlled trial. J Med Internet Res. 2014 Apr 4;16(4):e99. doi: 10.2196/jmir.3269. PMID 24705022
- See also: research group site web — http://calite.umh.es